CLINICAL TRIAL: NCT04136288
Title: Immediate and Short Term Efficacy of Low Intensity Shock Wave Therapy in the Management of Erectile Dysfunction Due to Mild - Moderate Cavernous Arterial Insufficiency
Brief Title: Low Intensity Shock Wave Therapy in the Management of Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gregory A. Broderick, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-001246
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Males with erectile dysfunction (ED) (Experimental): Males diagnosed with erectile dysfunction (ED) for over a year, but less than 5 years, will receive shock wave therapy via MoreNova device
  Interventions: Device: MoreNova

INTERVENTIONS:
Device: MoreNova — Shockwave therapy delivered to the genital area with low dose shocks

SUMMARY:
Researchers are evaluating the efficacy of low intensity shockwave therapy (LISWT) via MoreNova in the treatment of erectile dysfunction (ED).

DETAILED DESCRIPTION:
ED is broadly defined as the inability to achieve or maintain an erection sufficient for sexual intercourse or activity. Current treatment for ED consists of oral medications, intracavernosal injections and surgically placed penile prosthetics. In the literature this has been described as a Stepwise Approach, offering therapy beginning with the least invasive treatment option.

The goal of LISWT is to restore natural erections and / or improve responses to oral medications (first line therapy).

LISWT for ED is under evaluation in the USA. The European Association of Urology Guidelines on ED were recently updated to include LISWT for men with mild to moderate ED. The energy/pulse used in this application is approximately 10% of the energy used for disintegrating kidney stones; no serious side effects have been reported. Shock wave therapy for diabetic ulcers has recently been approved by the FDA.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his informed and signed written consent
* The patient is a male
* Between 40 to and including 55 years of age
* The patient has ED for longer than 1 year but less than 5 years.
* The patient is PDE5i responsive, meaning he is able to achieve and maintain an erection under the effect of the maximal dosage of PDE5i
* IIEF-EF Domain score of 17-20
* Evidence Based Criteria: Doppler Clinical Exam

Exclusion Criteria:

* The patient is participating in another study that may interfere with the results or conclusions of this study
* History of radical prostatectomy or extensive pelvic surgery
* Past radiation therapy of the pelvic region within 12 months prior to enrollment
* Recovering from cancer within 12 months prior to enrollment
* Neurological disease which effects erectile function
* Psychiatric disease which effects erectile function
* The patient is taking blood thinners
* History of Diabetes Mellitus
* History of Coronary Artery Disease
* Evidence Based Criteria: Doppler Clinical Exam
* Severe erectile dysfunction with IIEF-EF domain score < 16

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Broderick, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Males With Erectile Dysfunction (ED)
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Males With Erectile Dysfunction (ED)
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 51 [45 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 31.64 [24.29 to 41]

OUTCOME MEASURES:

1. Primary Outcome: Change in Right Resistive Index
Description: Resistive Index (RI) is a measure of resistance to blood flow within the right penile arteries.
  Measured using a Color Duplex Doppler Ultrasound (CDDU) measured in cm/second
  Elevated values are associated with a poorer prognosis. Lower values are associated with a better prognosis.
Time Frame: Treatment 6 Final Shockwave treatment (pre-procedure, intra-procedure, post procedure) approximately 1 hour
Measure: Mean (Full Range); unit: cm/second
Arm/Group | Males With Erectile Dysfunction (ED)
Number analyzed (Participants) | 6
cm/second | 75.67 [64 to 100]

2. Primary Outcome: Change in Right Peak Systolic Velocity
Description: Peak systolic velocity (PSV): The maximum velocity of blood flow during erection.
  Measured using a Color Duplex Doppler Ultrasound (CDDU) measured in cm/second
  A PSV higher than 35 cm/sec is regarded as normal, a 25-35 cm/sec may indicate moderate-to-mean arterial damage, and a PSV lower than 25 may indicate the presence of severe arteriopathy.
Time Frame: Treatment 6 Final Shockwave treatment (pre-procedure, intra-procedure, post procedure) approximately 1 hour
Measure: Mean (Full Range); unit: cm/second
Arm/Group | Males With Erectile Dysfunction (ED)
Number analyzed (Participants) | 6
cm/second | 16.27 [3.7 to 50.5]

3. Primary Outcome: Change in Right Diastolic Velocity
Description: Diastolic Velocity (DV) represents the velocity of right-side blood flow during the resting phase of the cardiac cycle. A DV less than 5 cm/s is considered normal (better). A DV less considered abnormal (worse).
  Measured using a Color Duplex Doppler Ultrasound (CDDU) measured in cm/second
Time Frame: Treatment 6 Final Shockwave treatment (pre-procedure, intra-procedure, post procedure) approximately 1 hour
Measure: Mean (Full Range); unit: cm/second
Arm/Group | Males With Erectile Dysfunction (ED)
Number analyzed (Participants) | 6
cm/second | 13.42 [0 to 26.7]

4. Primary Outcome: Erection Hardness Score (EHS)
Description: Measured using a self-reported Erection Hardness Score (EHS) scale options from 0 (minimum) to 4 (maximum).
  0- Penis does not enlarge, 1- Penis is larger but not hard, 2- Penis is hard but not hard enough for penetration, 3- Penis is hard enough for penetration but not completely hard, or 4-Penis is completely hard and fully rigid.
  A lower score indicates a worse outcome. A higher score indicates a better outcome.
Time Frame: Treatment 6 Final Shockwave treatment (pre-procedure, intra-procedure, post procedure) approximately 1 hour
Measure: Number; unit: participants
Arm/Group | Males With Erectile Dysfunction (ED)
Number analyzed (Participants) | 6
participants
  Number of participants who answered 0 on scale. | 0
  Number of participants who answered 1 on scale. | 1
  Number of participants who answered 2 on scale. | 1
  Number of participants who answered 3 on scale. | 4
  Number of participants who answered 4 on scale. | 0

5. Primary Outcome: International Index of Erectile Function (IIEF - EF) Questionnaire
Description: Measured using a self-reported International Index of Erectile Function questionnaire (IIEF - EF) consisting of 6 questions regarding the participants erectile function for the past 4 weeks. The questionnaire utilizes a scale of 0 (minimum) to 5 (maximum).
  A lower score indicates a worse outcome. A higher score indicates a better outcome.
  Questions 1-2 scale: 0=No sexual activity, 1= Almost never/never, 2= A few times (much less than half the time),3= Sometimes (about half the time), 4= Most times (much more than half the time),5= Almost always/always
  Questions 3-4 scale: 0=Did not attempt, 1=Almost never/never, 2= A few times (much less than half the time), 3= Sometimes (about half the time), 4= Most times (much more than half the time), 5= Almost always/always
  Question 5 scale:0=Did not attempt intercourse,1= Extremely difficult, 2=Very Difficult, 3=Difficult, 4= Slightly Difficult, 5= No Difficult
  Question 6 scale: 1= Very low, 2=Low, 3=Moderate, 4=High, 5= Very high
Time Frame: Treatment 6 Final Shockwave treatment (pre-procedure, intra-procedure, post procedure) approximately 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Males With Erectile Dysfunction (ED)
Number analyzed (Participants) | 6
Participants
  How often were you able to get an erection during sexual activity?: 0 | 1
  How often were you able to get an erection during sexual activity?: 1 | 1
  How often were you able to get an erection during sexual activity?: 2 | 1
  How often were you able to get an erection during sexual activity?: 3 | 1
  How often were you able to get an erection during sexual activity?: 4 | 2
  How often were you able to get an erection during sexual activity?: 5 | 0
  When you had erections with stimulation, how often were your erections hard enough for penetration?: 0 | 1
  When you had erections with stimulation, how often were your erections hard enough for penetration?: 1 | 2
  When you had erections with stimulation, how often were your erections hard enough for penetration?: 2 | 0
  When you had erections with stimulation, how often were your erections hard enough for penetration?: 3 | 1
  When you had erections with stimulation, how often were your erections hard enough for penetration?: 4 | 0
  When you had erections with stimulation, how often were your erections hard enough for penetration?: 5 | 2
  When you attempted sexual intercourse, how often were you able to penetrate your partner?: 0 | 2
  When you attempted sexual intercourse, how often were you able to penetrate your partner?: 1 | 1
  When you attempted sexual intercourse, how often were you able to penetrate your partner?: 2 | 0
  When you attempted sexual intercourse, how often were you able to penetrate your partner?: 3 | 1
  When you attempted sexual intercourse, how often were you able to penetrate your partner?: 4 | 1
  When you attempted sexual intercourse, how often were you able to penetrate your partner?: 5 | 1
  During intercourse,how often were you able to maintain your erection after you entered your partner?: 0 | 2
  During intercourse,how often were you able to maintain your erection after you entered your partner?: 1 | 1
  During intercourse,how often were you able to maintain your erection after you entered your partner?: 2 | 1
  During intercourse,how often were you able to maintain your erection after you entered your partner?: 3 | 1
  During intercourse,how often were you able to maintain your erection after you entered your partner?: 4 | 1
  During intercourse,how often were you able to maintain your erection after you entered your partner?: 5 | 0
  During intercourse, how difficult was it to maintain your erection to completion of intercourse?: 0 | 2
  During intercourse, how difficult was it to maintain your erection to completion of intercourse?: 1 | 1
  During intercourse, how difficult was it to maintain your erection to completion of intercourse?: 2 | 1
  During intercourse, how difficult was it to maintain your erection to completion of intercourse?: 3 | 1
  During intercourse, how difficult was it to maintain your erection to completion of intercourse?: 4 | 0
  During intercourse, how difficult was it to maintain your erection to completion of intercourse?: 5 | 1
  How would you rate your confidence that you could get and keep an erection?: 0 | 0
  How would you rate your confidence that you could get and keep an erection?: 1 | 2
  How would you rate your confidence that you could get and keep an erection?: 2 | 1
  How would you rate your confidence that you could get and keep an erection?: 3 | 3
  How would you rate your confidence that you could get and keep an erection?: 4 | 0
  How would you rate your confidence that you could get and keep an erection?: 5 | 0

6. Primary Outcome: Sexual Encounter Profile (SEP) Questionnaire
Description: Measured using a self-reported Sexual Encounter Profile (SEP) Questionnaire consisting of 2 questions. The questionnaire utilized Yes or No response options.
  No, indicates a worse outcome. Yes, indicates a better outcome.
Time Frame: Treatment 6 Final Shockwave treatment (pre-procedure, intra-procedure, post procedure) approximately 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Males With Erectile Dysfunction (ED)
Number analyzed (Participants) | 6
Participants
  Q2: Over the past 4 weeks, were you able to insert your penis into your partner's vagina.: Answered Yes | 3
  Q2: Over the past 4 weeks, were you able to insert your penis into your partner's vagina.: Answered No | 3
  Q3:Over the past 4 weeks, you had an erection last long enough to have successful intercourse.: Answered Yes | 2
  Q3:Over the past 4 weeks, you had an erection last long enough to have successful intercourse.: Answered No | 4

7. Primary Outcome: Global Assessment Questionnaire
Description: Measured using a self-reported Global Assessment Questionnaire consisting of 2 questions. The questionnaire utilized Yes or No response options.
  No, indicates a worse outcome. Yes, indicates a better outcome.
Time Frame: Treatment 6 Final Shockwave treatment (pre-procedure, intra-procedure, post procedure) approximately 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Males With Erectile Dysfunction (ED)
Number analyzed (Participants) | 6
Participants
  Q1: Over the past 4 week, has the treatment you have been taking improved your erectile function?: Answered Yes | 1
  Q1: Over the past 4 week, has the treatment you have been taking improved your erectile function?: Answered No | 5
  Q1: Over the past 4 week, has the treatment you have been taking improved your erectile function?: No response | 0
  Q2: Has the treatment improved your ability to engage in sexual activity over the past 4 weeks?: Answered Yes | 0
  Q2: Has the treatment improved your ability to engage in sexual activity over the past 4 weeks?: Answered No | 4
  Q2: Has the treatment improved your ability to engage in sexual activity over the past 4 weeks?: No response | 2

8. Primary Outcome: Change in Left Peak Systolic Velocity
Description: Measured using a Color Duplex Doppler Ultrasound (CDDU) measured in cm/second
  A Peak Systolic Velocity of 25-35 cm/s or higher is considered normal. This reflects the maximum velocity of blood flow during erection.
Time Frame: Treatment 6 Final Shockwave treatment (pre-procedure, intra-procedure, post procedure) approximately 1 hour
Measure: Mean (Full Range); unit: cm/second
Arm/Group | Males With Erectile Dysfunction (ED)
Number analyzed (Participants) | 6
cm/second | 26.63 [4.2 to 85.9]

9. Primary Outcome: Change in Left Diastolic Velocity
Description: Diastolic Velocity (DV) represents the velocity of left-side blood flow during the resting phase of the cardiac cycle. A DV less than 5 cm/s is considered normal (better). A DV less considered abnormal (worse).
  Measured using a Color Duplex Doppler Ultrasound (CDDU) measured in cm/second
Time Frame: Treatment 6 Final Shockwave treatment (pre-procedure, intra-procedure, post procedure) approximately 1 hour
Measure: Mean (Full Range); unit: cm/second
Arm/Group | Males With Erectile Dysfunction (ED)
Number analyzed (Participants) | 6
cm/second | 14.72 [7.2 to 32]

10. Primary Outcome: Left Resistive Index
Description: Resistive Index (RI) is a measure of resistance to blood flow within the left penile arteries.
  Measured Left Resistive Index using a Color Duplex Doppler Ultrasound (CDDU) measured in cm/second
  Elevated values are associated with poorer prognosis. Lower values are associated with a better prognosis.
Time Frame: Treatment 6 Final Shockwave treatment (pre-procedure, intra-procedure, post procedure) approximately 1 hour
Measure: Mean (Full Range); unit: cm/second
Arm/Group | Males With Erectile Dysfunction (ED)
Number analyzed (Participants) | 6
cm/second | 73.5 [60 to 84]

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Males With Erectile Dysfunction (ED)
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
The Covid-19 Pandemic was a limitation during the trial. The pandemic interfered with recruitment and follow-up of study subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT04136288/Prot_000.pdf